CLINICAL TRIAL: NCT05764421
Title: Motor-cognitive Interventions Are Effective in Improving Cognitive Function in Older Adults With Mild Cognitive impairment--a Chinese Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinxuan Cheng (Other)
Responsible Party: Sponsor-Investigator, Jinxuan Cheng, Principal Investigator, Qingdao University
Organization: Qingdao University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JCheng
Record Dates: First submitted 2023-02-27; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: MCI
Keywords: motor-cognitive intervention; older adults; cognitive ability; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention groups (Experimental): The experimental group received a uniform exercise - cognitive intervention at a community health centre or a geriatric activity station. The intervention lasted for a total of 12 weeks at a frequency of once every fortnight, with each intervention lasting 60-90 minutes. At the end of the intervention, the participants were followed up by the researchers for a total of 12 weeks, at a frequency of once every fortnight.
  The intervention consisted of physical-motor activities as well as integrated cognitive training.
  Interventions: Behavioral: motor-cognitive intervention
- control group (No Intervention): Participants in the control group did not undergo any intervention and kept their old lifestyle unchanged. The control group was asked to avoid cognitive training and exercise training beyond the routine throughout the investigation.

INTERVENTIONS:
Behavioral: motor-cognitive intervention — The intervention included physical activity and integrated cognitive training. The training was conducted in three sessions. The first session was a warm-up and wake-up preparation, in which participants massaged facial acupoints in a seated position to light music. In the middle phase of aerobic exercise, participants raised their legs in a standing position and performed mental exercises to fast-paced music. Session 1: tapping the five fingers of each hand in turn; Section 2: The thumb of both hands in turn to tap the rest of the fingers; Third section: hands five fingers cross fist; Section 4: The five fingers of both hands are stretched out in turn, and then retracted in turn. The final session was a relaxation session in which participants performed inspiratory and expiratory exercises to light music. The integrated cognitive training consisted of 15 minutes of attention training, 15 minutes of memory training, and 15 minutes of executive function training.
  Arms: intervention groups

SUMMARY:
Mild cognitive impairment (MCI) is a syndrome that occurs in the preclinical stage of Alzheimer, and early intervention can be effective in preventing Alzheimer, but further research is needed on intervention methods. In order to identify interventions that are more suitable for Chinese characteristics and to investigate the effects of a motor-cognitive intervention on the cognitive function of older adults with MCI, investigators screened 103 community-dwelling older adults with MCI aged 65 years and older in Qingdao, Shandong, China, and divided them into an intervention group and a control group, and administered a motor-cognitive intervention to the intervention group for 12 weeks. Investigators assessed the cognitive abilities of MCI participants using the Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA). There were no demographic differences between the intervention and control groups. Investigators found that the cognitive abilities of the intervention group were significantly improved at the end of the intervention as well as at the end of the follow-up compared to the control group. The results of the current study suggest that the motor-cognitive intervention investigators used significantly improved cognitive function in older adults with MCI and was easy for older adults to master, and that it was a good intervention for cognitive function in older adults with MCI in the Chinese community.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old;
* The screening results were mild cognitive impairment;
* Those who have the ability to walk independently or use auxiliary tools and can ·Communicate with each other normally;
* Informed consent, willing to participate in the researcher.

Exclusion Criteria:

* People with mental disorders;
* Patients with serious organ diseases, such as kidney and heart failure;
* People with mobility disabilities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Generalized estimating equations for the two groups of MMSE scores at three time points | 2020.8-2021.2
  The Shapiro-Wilk test was used to assess the normality of the data and found that the MMSE scores of the two groups of MCI participants were not normally distributed at all three time points, so we used medians and quartiles to describe the data. Generalized estimating equations were used to analyze the trends in MMSE scores at each time point for both groups. As seen in Table 4, the MMSE scores in the intervention group showed an increasing trend over time compared to the control group. There was a significant time effect (χ² = 27.259, p < 0.001) and a significant group effect (χ² = 21.267, p < 0.001) for the MMSE scores of the two groups. This indicates that the intervention used in this study was effective in improving the cognitive level of MCI patients in the intervention group. In order to visualize the trend in MMSE scores, a line graph was used to represent the change.
Between-group comparison of the MMSE scores of the two study groups at different time points | 2020.8-2021.2
  At different time points, the MMSE scores of the two study groups were not normally distributed, therefore, the between-group differences in the MMSE scores of the two study groups at the three time points were statistically analyzed using a two independent samples non-parametric rank sum test. The results showed a significant difference in MMSE scores between the two groups of participants at the end of the intervention (Z = 5.406, p < 0.001). At the end of follow-up, there was a significant difference in MMSE scores between the two groups of participants (Z = 5.403, p < 0.001).
Intra-group comparison of MMSE scores between the two groups | 2020.8-2021.2
  As the MMSE scores of MCI older adults in both the intervention and control groups were not normally distributed at all three time points, a paired rank sum test was used to compare the change in MMSE scores between the two groups of participants before and after the intervention. The results showed that MMSE scores in the intervention group were significantly higher at the end of the intervention compared to the initial level (Z = -4.287, p < 0.001). MMSE scores in the intervention group were significantly higher at the end of follow-up compared to initial levels (Z = -4.251, p < 0.001).
Generalized estimating equations for MoCA scores for two groups of older people at three time points | 2020.8-2021.2
  The MoCA scores of the two groups of MCI older adults were not normally distributed at all three time points, so generalised estimating equations were used to analyze the trends in the MoCA scores of the two groups at each time point. As seen in Table 7, there was a significant upward trend in MoCA scores over time in the intervention group compared to the control group. There was a significant time effect (χ² = 46.922, p < 0.001) and a significant group effect (χ² = 60.992, p < 0.001) for the MoCA scores of the participants in both groups. This indicates that the intervention method used in this study was effective in improving the cognitive level of MCI patients in the intervention group. To visualize the trend of MoCA scores, a line graph was used to represent the trend.
Intergroup comparison of MoCA scores between the two study groups | 2020.8-2021.2
  The MoCA scores of the two study groups were not normally distributed at different time points, therefore, the between-group differences in the MoCA scores of the two study groups before the intervention, at the end of the intervention and at the end of follow-up were statistically analysed using a two independent samples non-parametric rank sum test. The results showed that the difference in MoCA scores between the two groups of participants at the end of the intervention was significant (Z = 6.108, p < 0.001). At the end of follow-up, there was a significant difference in MoCA scores between the two groups of participants (Z = 6.215, p < 0.001).
Intra-group comparison of MoCA scores between the two groups of older people | 2020.8-2021.2
  As the MoCA scores of MCI older adults in both the intervention and control groups were not normally distributed at the three time points, a paired rank sum test was used to compare the change in MoCA scores of the two groups of older adults before and after the intervention. The results showed that MoCA scores in the intervention group were significantly higher at the end of the intervention compared to the initial level (Z = -5.539, p < 0.001). MoCA scores in the intervention group were significantly higher at the end of follow-up compared to initial levels (Z = -5.330, p < 0.001).

CONTACTS AND LOCATIONS:
Locations (1):
- Jinxuan Cheng, Qingdao, Shandong, China